CLINICAL TRIAL: NCT07176936
Title: Noninvasive Vagus Nerve Stimulation for Improved Speech in Noise Perception
Brief Title: Improving Speech in Noise Using Noninvasive Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202500139; RH240016 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury; Hearing Loss
MeSH Terms: conditions — Brain Injuries, Traumatic; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment A vs Treatment B (Other): Participants will receive the stimulation at location A and then receive stimulation at location B, both on the outer ear.
  Interventions: Device: Cymba Conchae stimulation; Device: Earlobe stimulation
- Treatment B then Treatment A (Other): Participants will receive the stimulation at location B and then receive stimulation at location A, both on the outer ear.
  Interventions: Device: Cymba Conchae stimulation; Device: Earlobe stimulation

INTERVENTIONS:
Device: Cymba Conchae stimulation — Electrical stimulation applied to the cymba conchae region of the outer ear
  Other Names: Treatment A
Device: Earlobe stimulation — Electrical stimulation applied to the earlobe region of the outer ear
  Other Names: Treatment B

SUMMARY:
Traumatic brain injury, a common injury in military service personnel, often leads to poor processing of speech in noisy environments. The goal of the current study is to better understand the brain basis for this difficulty and evaluate a new approach to improving speech in noise perception.

ELIGIBILITY:
Inclusion Criteria:

* 25-55 years old
* Proficiency in English
* TBI group: history of traumatic brain injury by blast or physical trauma
* Normal hearing group: no history of traumatic brain injury

Exclusion Criteria:

* Other neurological diseases or related conditions will be excluded (e.g., large vessel stroke, seizures). We will exclude patients with severe medical diseases that may be associated with impaired cognition (e.g., heart failure, dialysis dependent kidney disease, brain cancer). Further, psychiatric diseases that are unlikely to be related to trauma will be excluded (e.g., schizophrenia).

Patients with histories of severe psychiatric disease prior to trauma exposure will be excluded.

* Current illicit or prescription drug abuse (within the last two months)
* Any taVNS contraindication, including but not limited to the presence of unremovable metal in the left ear, known heart conditions, medications that influence neurotransmitters thought to be critical for vagus nerve stimulation (norepinephrine, acetylcholine, and serotonin), or implanted medical devices such as a pacemaker.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility | From enrollment to the end of treatment is between 2 days and 2 weeks.
  quantify attrition as well as frequency and severity of adverse events

SECONDARY OUTCOMES:
Speech in Noise performance | Baseline and one week
  Percent correct on a speech in noise perception task when receiving Treatment A compared to Treatment B
Brain response patterns | Baseline and one week
  Pattern of brain response while listening to speech in background noise while receiving Treatment A compared to Treatment B

CONTACTS AND LOCATIONS:
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the time of data publication
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared at the time of publication and will be available indefinitely
Access Criteria: Data and protocols will be shared openly.